CLINICAL TRIAL: NCT02364336
Title: Mechanisms Associated With Favorable Response to Peginterferon-Alpha Add-on Therapy Following Long-term Nucleos(t)Ide Analogue Treatment in Patients With Chronic Hepatitis B
Brief Title: Add-on Peginterferon Following Nucleos(t)Ide Analogue Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150082; 15-DK-0082 (Other: NIDDK/NIH)
Record Dates: First submitted 2015-02-14; First posted 2015-02-18 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-05-21

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (2):
- HBeAg positive (Experimental): Patients who have been treated with one or more nucleos(t)ides for at least 192 weeks who have known serum HBsAg and HBeAg positivity
  Interventions: Drug: Peginterferon alfa-2a
- HBeAg negative (Experimental): Patients who have been treated with one or more nucleos(t)ides for at least 192 weeks who have known serum HBsAg positivity and HBeAg negativity
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a

SUMMARY:
Background:

- Chronic hepatitis B is caused by a virus that infects the liver. Cure is not possible but the virus can be controlled with the use of antiviral medicines,. Researchers think that adding a second antiviral medicine might help.

Objective:

- To understand how peginterferon might help treat people with chronic hepatitis B. Also, to see if peginterferon is safe to use with other antiviral medications.

Eligibility:

- Adults age 18 and older who have chronic hepatitis B and had therapy with 1 or more oral medicines for hepatitis B for at least 4 years.

Design:

* Participants will be screened with physical exam and medical history. They will complete health questionnaires about their levels of fatigue and pain. They will have blood and urine tests. They may have an eye exam.
* Participants also will have a Fibroscan. A test to measure how stiff your liver is.
* Eligible participants will have a liver biopsy. Blood will be drawn.
* Participants will be admitted to the NIH Clinical Center. They will be injected with the study drug. Then they will have a second liver biopsy. They will be discharged 24 hours later.
* Participants will give themselves study drug injections under the skin weekly for 24 weeks.
* Participants will have 5 clinic visits during the 24-week treatment period. Then they will have follow-up visits every 12 weeks for 48 weeks.
* During visits, participants may have a physical exam and medical history. They may have blood and urine tests. They may have a Fibroscan and complete questionnaires. At the final visit, they will also have a Fibroscan.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection is a leading cause of liver associated morbidity and mortality. Currently available first-line therapies for treatment of chronic hepatitis B include pegylated interferon-alpha and the nucleos(t)ide analogues (NUCs) entecavir and tenofovir. These were shown to effectively suppress viral replication, but their ability to induce durable off-treatment response is limited to a small subset of patients. Combination treatment with peginterferon and NUCs has been attempted in several randomized controlled trials, with no apparent advantage over either agent given alone. In these studies however, treatment with peginterferon was initiated either simultaneously or shortly after NUCs administration. The efficacy of peginterferon following long-term viral suppression with NUCs was only tested in one small pilot study, nevertheless showing 60% hepatitis B s antigen (HBsAg) loss rate.

The underlying mechanisms responsible for improved efficacy of peginterferon in this setting are unknown and warrant further investigation. In this single arm study we propose to evaluate the efficacy and mechanisms associated with response to peginterferon add-on therapy following a minimum of 192 weeks of viral suppression induced by NUCs in a group of chronic HBV infected patients. Sixty patients with either hepatitis B e antigen (HBeAg) positive (n=30) or negative (n=30) chronic HBV infection will be enrolled to this study. After medical evaluation and pretreatment liver biopsy, treatment with subcutaneous injections of pegylated interferon alpha-2a 180 g per week will be given for a total of 24 weeks, followed by an off-treatment evaluation period of 48 weeks. A second liver biopsy will be performed six hours following the first peginterferon injection. Primary end-point for this study will be the change in interferon-stimulated-genes response before and after first interferon injection in responders versus non-responders to treatment. The responsiveness to IFN-based therapy of treatment responders vs nonresponders will additionally be evaluated by studying intrahepatic and peripheral blood natural killer cells. The study will also assess HBeAg and HBsAg loss and seroconversion rates in comparison to historical controls treated with either peginterferon or NUCs monotherapy. Finally, we will assess whether treatment responders develop an HBV-specific T cell response similar in quantity and quality to that of patients who spontaneously resolve HBV infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria: HBeAg positive group

1. Age >18 years and older, male or female.
2. Known serum HBsAg and HBeAg positivity at the time of screening.
3. Ongoing treatment with one or more NUCs for at least 192 weeks before study entry. Subjects may have a brief interruption of treatment for medical reasons (e.g. breast feeding) not to exceed 8 weeks and none within the 48 weeks before study entry.
4. HBV DNA levels <100 IU/mL, measured at least 12 months prior to, and upon enrollment to the study.
5. ALT level less than or equal to 2 ULN based on at least two determinations taken at least one month apart during the 24 weeks before study entry with the second being at time of screening
6. Written informed consent

Inclusion criteria: HBeAg negative group

1. Age >18 years and older, male or female.
2. Known serum HBsAg positivity and HBeAg negativity at the time of screening.
3. Ongoing treatment with one or more NUCs for at least 192 weeks before study entry. Subjects may have a brief interruption of treatment for medical reasons (e.g. breast feeding) not to exceed 8 weeks and none within the 48 weeks before study entry.
4. HBV DNA levels <100 IU/mL, measured at least 12 months prior to, and upon enrollment to the study
5. ALT level less than or equal to 2 ULN based on at least two determinations taken at least one month apart during the 24 weeks before study entry with the second being at time of screening
6. Written informed consent

EXCLUSION CRITERIA:

Exclusion criteria (for both eAg positive and negative patients)

1. Co-infection with HDV as defined by the presence of anti-HDV in serum and/or HDV antigen in the liver.
2. Co-infection with HCV as defined by the presence of HCV RNA in serum.
3. Co-infection with HIV as defined by the presence of anti-HIV in serum.
4. Decompensated liver disease as defined by serum bilirubin >2.5 mg/dL (with direct bilirubin > 0.5 mg/dL), prothrombin time of greater than 2 seconds prolonged, a serum albumin of less than 3 g/dL, or a history of ascites, variceal bleeding or hepatic encephalopathy.
5. Presence of other causes of liver disease, (i.e. hemochromatosis, Wilson disease, alcoholic liver disease, severe nonalcoholic steatohepatitis defined as the presence of marked ballooning injury on liver biopsy, alpha-1-anti-trypsin deficiency).
6. A history of organ transplantation or in the absence of organ transplantation, any immunosuppressive therapy requiring the use of more than 5 mg of prednisone (or its equivalent) daily.
7. Significant systemic illness other than liver diseases including congestive heart failure, renal failure, chronic pancreatitis and diabetes mellitus with poor control, that in the opinion of the investigator may interfere with therapy.
8. Pregnancy or inability to practice contraception in patients capable of bearing or fathering children
9. Lactating women.
10. Hepatocellular carcinoma (HCC), or the presence of a mass on imaging studies of the liver that is suggestive of HCC, or an alpha-fetoprotein level of greater than 500 ng/mL.
11. eGFR < 50 ml/min, serum creatinine > 1.3 mg/dl or urine protein >1 gram/24-hours
12. History of hypersensitivity to pegylated interferon-alpha
13. Platelet count <70 mm(3)/dL
14. Hgb <12 g/dL for males and <11 g/dL for females
15. Active ethanol/drug abuse/psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, or personality disorder that, in the investigator s opinion, might interfere with participation in the study.
16. History of malignancy or treatment for a malignancy within the past 3 years (except adequately treated carcinoma in situ or basal cell carcinoma of the skin).
17. Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids or other immunosuppressive medications during the course of this study.
18. History of immune-mediated disease, or cerebrovascular, chronic pulmonary or cardiac disease associated with functional limitation, retinopathy, uncontrolled thyroid disease, poorly controlled diabetes or uncontrolled seizure disorder, as determined by a study physician.
19. Presence of conditions that, in the opinion of the investigators, would not allow the patient to be followed in the current study for at 1 year.
20. For subjects who interrupt therapy, documentation of a viral load >1,000 IU/ml while off therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-14; Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sadler AJ, Williams BR. Interferon-inducible antiviral effectors. Nat Rev Immunol. 2008 Jul;8(7):559-68. doi: 10.1038/nri2314. PMID 18575461
- [Background] Ouzan D, Penaranda G, Joly H, Khiri H, Pironti A, Halfon P. Add-on peg-interferon leads to loss of HBsAg in patients with HBeAg-negative chronic hepatitis and HBV DNA fully suppressed by long-term nucleotide analogs. J Clin Virol. 2013 Dec;58(4):713-7. doi: 10.1016/j.jcv.2013.09.020. Epub 2013 Sep 29. PMID 24183313
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0082.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening occurred after participant enrollment. 14 patients were enrolled. One participant failed screening, and 13 started treatment.
Period: Overall Study
Arm/Group | HBeAg Positive | HBeAg Negative
Started | 1 | 12
6 Hours Post First Peginterferon Inject | 1 | 12
End of Peginterferon Treatment | 1 | 11
24 Weeks After End of Peginterferon | 1 | 11
48 Weeks After End of Peginterferon | 1 | 10
Completed | 1 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HBeAg Positive | HBeAg Negative | Total
Number analyzed (Participants) | 1 | 12 | 13
Age, Continuous [Mean (Full Range); unit: years] | 35 [35 to 35] | 48 [24 to 69] | 48 [24 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 1 | 9 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 8 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Interferon-stimulated-gene (ISG) Expression
Description: Change in level of ISG expression before and after 1st peginterferon injection
Time Frame: 6 hours after first injection of peginterferon
Population: One patient with HBeAg positive had insufficient liver tissue to perform the RNASeq.
Measure: Mean (Standard Error); unit: log 2 fold change
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 1 | 12
log 2 fold change
  PPP1R3G: number analyzed (Participants) | 0 | 12
  PPP1R3G |  | -2.716 (0.628)
  ALAS1: number analyzed (Participants) | 0 | 12
  ALAS1 |  | 1.670 (0.416)
  INHBB: number analyzed (Participants) | 0 | 12
  INHBB |  | -2.20 (0.570)
  MMRN1: number analyzed (Participants) | 0 | 12
  MMRN1 |  | -1.597 (0.432)
  LYVE1: number analyzed (Participants) | 0 | 12
  LYVE1 |  | -1.184 (0.326)
  SLC8A1: number analyzed (Participants) | 0 | 12
  SLC8A1 |  | -1.382 (0.386)
  PPARGC1A: number analyzed (Participants) | 0 | 12
  PPARGC1A |  | -1.573 (0.443)
  NOTUM: number analyzed (Participants) | 0 | 12
  NOTUM |  | 0.870 (0.250)
  IGFBP3: number analyzed (Participants) | 0 | 12
  IGFBP3 |  | -0.723 (0.214)
  LTBP1: number analyzed (Participants) | 0 | 12
  LTBP1 |  | -0.548 (0.163)
  STARD5: number analyzed (Participants) | 0 | 12
  STARD5 |  | 1.798 (0.547)
  RTN4RL1: number analyzed (Participants) | 0 | 12
  RTN4RL1 |  | 1.808 (0.556)
  ZPR1: number analyzed (Participants) | 0 | 12
  ZPR1 |  | -0.972 (0.299)

2. Secondary Outcome: Hepatitis B e Antigen (HBeAg) Loss
Description: Proportion of HBeAg positive patients showing eAg loss at end of treatment, and 24 and 48 weeks off peginterferon treatment.
Time Frame: End of treatment, 24 weeks, and 48 weeks
Population: Outcome only applies to HBeAg positive patients
Measure: Count of Participants; unit: Participants
Arm/Group | HBeAg Positive
Number analyzed (Participants) | 1
Participants
  End of treatment | 0
  Week 24 post treatment | 0
  Week 48 post treatment | 0

3. Secondary Outcome: Hepatitis B s Antigen (HBsAg) Loss
Description: Proportion of HBsAg positive patients showing sAG loss at end of treatment and 24 and 48 weeks off peginterferon treatment
Time Frame: End of treatment, 24 weeks, and 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- HBeAg Negative: Patients who have been treated with one or more nucleos(t)ides for at least 192 weeks who have known serum HBsAg positivity and HBeAg negative
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 1 | 12
Participants
  End of treatment | 0 | 1
  Week 24 post treatment | 0 | 0
  Week 48 post treatment | 0 | 0

4. Secondary Outcome: Change in Natural Killer (NK) Cell Frequency
Description: NK cell frequency is calculated as 100*(NK cells)/(mononuclear cells). Changes are calculated by subtracting baseline from 6 hours after first peginterferon injection.
Time Frame: 6 hours after first injection of peginterferon and baseline
Population: One patient with HBeAg positive had insufficient liver tissue to obtain frequency and degranulation measurement in liver.
Measure: Mean (Standard Deviation); unit: percentage of mononuclear cells
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 1 | 12
percentage of mononuclear cells
  Blood baseline | 15.60 (NA) — There is only one patient and standard deviation cannot be obtained. | 11.82 (10.19)
  Blood 6 hours | 10.30 (NA) — There is only one patient and standard deviation cannot be obtained. | 13.74 (10.68)
  Blood change | -5.3 (NA) — There is only one patient and standard deviation cannot be obtained. | 1.92 (7.48)
  Liver baseline: number analyzed (Participants) | 0 | 12
  Liver baseline |  | 24.69 (6.26)
  Liver 6 hours: number analyzed (Participants) | 0 | 12
  Liver 6 hours |  | 24.78 (7.28)
  Liver change: number analyzed (Participants) | 0 | 12
  Liver change |  | 0.09 (4.08)

5. Secondary Outcome: Change in Natural Killer (NK) Cell Degranulation
Description: NK cell degranulation is calculated as 100*(degranulated NK cells)/(NK cells). Changes are calculated by subtracting baseline from 6 hours after first peginterferon injection.
Time Frame: 6 hours after first injection of peginterferon and baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % of NK cells
Arm/Group | HBeAg Positive | HBeAg Negative
Number analyzed (Participants) | 1 | 12
% of NK cells
  Blood baseline | 0.08 (NA) — There is only one patient and standard deviation cannot be obtained. | 0.64 (0.65)
  Blood 6 hours | 0.06 (NA) — There is only one patient and standard deviation cannot be obtained. | 0.52 (0.66)
  Blood change | -0.02 (NA) — There is only one patient and standard deviation cannot be obtained. | -0.12 (0.93)
  Liver baseline: number analyzed (Participants) | 0 | 12
  Liver baseline |  | 3.37 (1.46)
  Liver 6 hours: number analyzed (Participants) | 0 | 12
  Liver 6 hours |  | 4.87 (4.47)
  Liver change: number analyzed (Participants) | 0 | 12
  Liver change |  | 1.51 (5.08)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over three periods encompassing a total of 50 to 60 weeks. The first period was up to twelve weeks, from pre-treatment biopsy to start of peginterferon treatment. The second period was 24 weeks during treatment with peginterferon, and the third period was after completion of treatment with peginterferon.
Arm/Group | HBeAg Positive | HBeAg Negative
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/12
Other Adverse Events (participants affected / at risk) | 1/1 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBeAg Positive (N=1) | HBeAg Negative (N=12)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HBeAg Positive (N=1) | HBeAg Negative (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 | 5
Anorexia (Gastrointestinal disorders) | 1 | 9
Anxiety (Psychiatric disorders) | 0 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Biopsy Site Pain (Injury, poisoning and procedural complications) | 0 | 4
Blurred Vision (Eye disorders) | 0 | 5
Chills (General disorders) | 1 | 7
Constipation (Gastrointestinal disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Diarrhea (Gastrointestinal disorders) | 0 | 5
Dizziness (Nervous system disorders) | 0 | 8
Dry Mouth (Gastrointestinal disorders) | 0 | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 8
Fast or pounding heartbeat (Cardiac disorders) | 1 | 4
Fatigue (General disorders) | 1 | 12
Fever (General disorders) | 1 | 5
Urinary frequency (Renal and urinary disorders) | 1 | 7
hair loss (Skin and subcutaneous tissue disorders) | 0 | 5
headache (Nervous system disorders) | 1 | 11
insomnia (Psychiatric disorders) | 1 | 9
irritability (Psychiatric disorders) | 1 | 6
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 9
joint pain (Musculoskeletal and connective tissue disorders) | 1 | 6
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 11
nausea (Gastrointestinal disorders) | 1 | 6
rash (Skin and subcutaneous tissue disorders) | 0 | 4
melancholy (Psychiatric disorders) | 0 | 7
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 4
toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Weight loss (Investigations) | 1 | 8
irritation at injection site (Injury, poisoning and procedural complications) | 1 | 3
Indigestion (Gastrointestinal disorders) | 0 | 1
infection (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT02364336/Prot_SAP_000.pdf